CLINICAL TRIAL: NCT05193487
Title: Influence Of Computerized Intraosseous Anesthesia On Children's Behaviour In Comparison To Traditional Mandibular Nerve Block Technique: A Randomized Clinical Trial
Brief Title: Intraosseous Anesthesia Versus Mandibular Nerve Block in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mariem Wassel, Clinical assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDASU-Rec R102110
Record Dates: First submitted 2021-12-08; First posted 2022-01-18 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Dental Anaesthesia
Keywords: intra-osseous anesthesia; inferior alveolar nerve block

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inferior alveolar nerve block (Active Comparator): Conventional inferior alvoelar nerve block anaesthesia will be given using a traditional metal syringe
  Interventions: Other: inferior alveolar nerve block
- intra-osseous mandibular anaesthesia (Experimental): Computerized intraosseous anesthesia administration using the Quick Sleeper 5TM system (Dental Hi TecTM, Cholet, France)
  Interventions: Other: intra-osseous mandibular anaesthesia

INTERVENTIONS:
Other: inferior alveolar nerve block — inferior alveolar nerve block using Articaine 4% with 1/200000 Adrenaline and a traditional needle injection
  Arms: inferior alveolar nerve block
Other: intra-osseous mandibular anaesthesia — intra-osseous mandibular anaesthesia using Articaine 4% with 1/200000 Adrenaline and a special intra-osseous injection device
  Arms: intra-osseous mandibular anaesthesia

SUMMARY:
The aim of the current study is to compare a new computerized intra-osseous injection system to the conventional inferior alveolar nerve block in children

DETAILED DESCRIPTION:
Patients will be randomly allocated to one of the experimental groups.: Conventional (Inferior alveolar nerve block) and Computerized intraosseous anesthesia administration using the Quick Sleeper 5TM system (Dental Hi TecTM, Cholet, France). Both techniques will be performed by a single trained operator.

Articaine 4% with 1/200000 Adrenaline will be used for both techniques.

ELIGIBILITY:
Inclusion criteria

1. Children aging between 6-9 years with no history of previous local dental anesthesia experience.
2. American society of anesthesiologists score equal to or less than II
3. Lower 2nd primary molars requiring pulpotomy

Exclusion criteria:

1. American society of anesthesiologists Score more than II
2. Uncompliant, Uncooperative children
3. Children turning non-compliant during procedure
4. Patients taking analgesics and anti-inflammatory
5. Un-restorable teeth, teeth near exfoliation, teeth with gingival abscess/fistula, pathological mobility, pain on percussion, radiographic evidence of internal or external pathological root resorption, periapical/furcation radio-lucencies, widened periodontal membrane space.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Patient's level of cooperation | directly after anesthetic injection while providing the dental treatment
  The child behavior will be evaluated using the modified Venham scale (scores 0-5) where higher scores indicate uncooperative behavior

SECONDARY OUTCOMES:
Heart Rate | before injection, during injection and directly after injection.
  Heart Rate (physiological measure)
Anesthesia success or failure | directly after anesthetic injection while providing the dental treatment
  Completing the needed treatment will be recorded as anesthesia success while failure to complete pulpotomy due to pain will be recorded as anesthesia failure

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Zayed, lecturer, Principal Investigator — Faculty of Dentistry, Ain Shams University, Cairo, Eypt
Locations (1):
- Faculty of Dentistry, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Radwan MZ, Wassel MO, El Geleel OA, Elghazawy RK. Influence of computerized intraosseous anesthesia compared with traditional mandibular nerve block on children's behavior: A randomized clinical trial. Int J Paediatr Dent. 2025 Mar;35(2):281-288. doi: 10.1111/ipd.13231. Epub 2024 Jun 24. PMID 38923102